CLINICAL TRIAL: NCT05441124
Title: The Effect of Web-based Mindfulness-Based Stress Reduction Program on Prenatal Comfort and Fetal Anxiety Levels in Pregnants
Brief Title: The Effect of Web-based Mindfulness-based Stress Reduction Program on Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amasya University (Other)
Responsible Party: Principal Investigator, Emine Akca, Assist. Prof. Dr. in the Amasya University Midwifery Department, Amasya University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Amasya Uni
Record Dates: First submitted 2022-06-28; First posted 2022-07-01 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Anxiety; Pregnancy Related
Keywords: Prenatal Comfort; MBSR
MeSH Terms: conditions — Anxiety Disorders | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfullness Based Stress Reduction (Experimental): Mindfullness Based Stress Reduction (MBSR) therapy
  Interventions: Behavioral: Mindfullness Based Stress Reduction (MBSR) intervention
- Control (No Intervention): Control

INTERVENTIONS:
Behavioral: Mindfullness Based Stress Reduction (MBSR) intervention — Mindfullness Based Stress Reduction (MBSR) intervention: Monitoring stress and anxiety levels with mindfulness program
  Arms: Mindfullness Based Stress Reduction

SUMMARY:
Pregnancy is a period in which physiological and psychological changes are experienced and discomforts related to these changes are observed, and comfort is affected for the pregnant. However, fetal health concern refers to the concern of the expectant mother about the health of her developing fetus. Mindfulness is a non-judgmental and accepting focus of one's attention on what is happening right now. A total of 96 pregnant women (48 experimental, 48 control) are planned to be included in the study. Data will be collected with the "Personal Description Form", "Prenatal Comfort Scale (PCS)" and "Fetal Health Anxiety Inventory (FHAI)". In the study, a stress reduction program (MBSR) based on mindfulness will be applied by the researcher to the pregnant women in the experimental group.

DETAILED DESCRIPTION:
Women experience intense physiological, psychological and social changes during pregnancy and postpartum period. Pregnancy and postpartum period can be a difficult process for some women due to biological and environmental factors. Mindfulness-based approaches have been used in solving both physical and mental problems in pregnant women and very positive results have been obtained. The aim of this study, which is carried out to determine the effect of mindfulness on prenatal comfort and fetal anxiety levels in pregnant women, is aimed at creating intervention programs compatible with the antenatal period and contributing to the improvement of pregnancy outcomes. A total of 96 pregnant women (48 experimental, 48 control) are planned to be included in the study. Data will be collected with the "Personal Description Form", "Prenatal Comfort Scale (PCS)" and "Fetal Health Anxiety Inventory (FHAI)". In the study, a stress reduction program (MBSR) based on mindfulness will be applied by the researcher to the pregnant women in the

ELIGIBILITY:
Inclusion Criteria:

* Not having any diagnosed psychiatric disease,
* Literate,
* Using a smart phone,
* With internet access
* Having a headset accessory for phone calls,
* Pregnant women who voluntarily agreed to participate in the study

Exclusion Criteria:

* Filling in the questionnaire form incompletely,
* Pregnant women with communication barriers and mental disabilities

Ages: 15 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Pregnant
Enrollment: 89 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Prenatal Comfort Scale | At the end of the 2 months
  The minimum score that can be obtained from the scale is "0", the maximum score is "75", and as the score obtained from the scale increases, prenatal comfort levels also increase.
Fetal Health Anxiety Inventory | At the end of the 2 months
  The minimum score that can be obtained from the scale is "0", the maximum score is "42", and as the score obtained from the scale increases, fetal health anxiety levels also increase.

CONTACTS AND LOCATIONS:
Locations (1):
- Amasya University, Amasya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No